CLINICAL TRIAL: NCT07379398
Title: A Single-center, Single-arm Clinical Study on the Efficacy and Safety of Iparomlimab and Tuvonralimab Injection Combined With SBRT in Patients With Early-Stage Non-Small Cell Lung Cancer
Brief Title: Iparomlimab and Tuvonralimab Injection Combined With SBRT in Patients With Early-Stage Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251143A
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
Keywords: lparomlimab and Tuvonralimab Injection; SBRT; early-stage
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lparomlimab and Tuvonralimab Injection in Combination with SBRT (Experimental): lparomlimab and Tuvonralimab Injection in Combination with SBRT
  Interventions: Drug: lparomlimab and Tuvonralimab Injection in Combination with SBRT

INTERVENTIONS:
Drug: lparomlimab and Tuvonralimab Injection in Combination with SBRT — lparomlimab and Tuvonralimab Injection: 5 mg/kg, administered every 3 weeks (q3w). The first dose should be given within one week after the initial SBRT fraction. The treatment duration is one year.
  SBRT: 50 Gy in 4 fractions or 70 Gy in 10 fractions, to be completed within 1-2 weeks.

SUMMARY:
Major objectives to evaluate the efficacy and safety of lparomlimab and Tuvonralimab Injection ((QL1706, an Anti-PD-1/CTLA-4 Combined Antibody)) combined with SBRT in patients with early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
This single-arm, single-center clinical study aims to evaluate the efficacy and safety of lparomlimab and Tuvonralimab Injection ((QL1706, an Anti-PD-1/CTLA-4 Combined Antibody)) combined with SBRT in patients with early-stage non-small cell lung cancer. This study consists of three phases: screening, treatment, and follow-up.Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent form for this study;
* Age ≥ 18 years;
* ECOG performance status of 0-1;
* Histologically confirmed non-small cell lung cancer, meeting AJCC 8th edition Stage IA-IB (tumor size ≤ 4cm, N0M0), Stage IIA (≤5cm, N0M0), or Stage IIB (>5cm and ≤7cm, N0M0);
* At least one repeatable measurable lesion at baseline (according to RECIST 1.1 criteria);
* Function of vital organs within 7 days prior to initial treatment meets the following requirements (use of any blood components or colony-stimulating factors within 14 days prior to enrollment is not allowed): Hemoglobin (Hb) ≥ 90 g/L; White Blood Cell (WBC) count ≥ 3.5 × 10^9/L; Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L; Platelets (PLT) ≥ 80 × 10^9/L; Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × Upper Limit of Normal (ULN); if liver metastases are present, AST and ALT ≤ 5 × ULN; Total Bilirubin (TBIL) ≤ 1.5 × ULN; Blood Urea Nitrogen (BUN) and Creatinine (Cr) ≤ 1.5 × ULN (and Creatinine Clearance (CCr) ≥ 50 mL/min); Left Ventricular Ejection Fraction (LVEF) ≥ 50%; QT interval corrected by Fridericia's formula (QTcF) < 470 milliseconds;
* Eligible patients of childbearing potential must agree to use a reliable method of contraception together with their partner during the trial period and for at least 180 days after the last dose of the study drug.

Exclusion Criteria:

* Inability to comply with the research protocol or study procedures.
* Previous receipt of any treatment, including chemotherapy or radiotherapy, for the currently diagnosed lung cancer.
* Patients with positive driver gene mutations such as EGFR, ALK, or ROS1.
* History of allergy or hypersensitivity to the investigational drug(s) or any of their excipients, or a history of atopy.
* Presence of active pulmonary tuberculosis, radiation pneumonitis, drug-induced pneumonitis, or other diseases, symptoms, or signs indicating severe pulmonary impairment during the screening period.
* Concurrent severe cardiovascular or cerebrovascular diseases.
* Receipt of broad-spectrum antibiotic therapy via any route within 30 days prior to the first dose.
* Positive anti-HIV test; positive Hepatitis B surface antigen (HBsAg) with HBV-DNA above the upper limit of normal (ULN); active Hepatitis C virus (HCV) infection.
* Evident bleeding tendency or other significant evidence of coagulation disorders.
* Current interstitial pneumonia or interstitial lung disease, or a prior history of interstitial pneumonia or interstitial lung disease requiring corticosteroid treatment; or other conditions such as pulmonary fibrosis or organizing pneumonia that may interfere with the assessment and management of immune-related pulmonary toxicity.
* Clinically symptomatic moderate or severe ascites requiring therapeutic paracentesis or drainage (except for cases with only minimal ascites visible on imaging without clinical symptoms), or uncontrolled or moderate-to-large pleural effusion or pericardial effusion.
* Ongoing systemic corticosteroid therapy or other immunosuppressive agents within 14 days prior to the first dose, or use of immunostimulants (including but not limited to interferon or interleukin-2) within 4 weeks prior.
* Diagnosis of other malignancies within 5 years prior to enrollment, except for radically resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix.
* Active autoimmune disease or a history of autoimmune disease within 4 weeks prior to enrollment.
* Patients deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
1-year EFS | up to 12 month

SECONDARY OUTCOMES:
Objective response rate | up to 12 month
  the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment.
Overall survival | up to 36 month
  OS was defined as the time from the first dose of study drug to death due to any cause.
Adverse Events | up to 36 month
  An AE was defined as any untoward medical occurrence in a pharmaceutical productwhich does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No